CLINICAL TRIAL: NCT07183475
Title: Amendment to the Study "Prospective, Multicenter Investigation of Clinical Rehabilitation and Everyday Recovery Following Knee Joint Endoprosthetic Replacement" With Additional Return-to-sports-testing at One Participating Center
Brief Title: Return to Sports After Knee Arthroplasty
Acronym: RTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-687_1-S-CB
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthristis; Arthroplasty Replacement, Knee
Keywords: return to sports; knee oteoarthritis; knee arthroplasty

STUDY DESIGN:
Intervention Model Description: single-center, prospective pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RTS (Experimental): Return-to-sports-tested patients
  Interventions: Diagnostic Test: Return to sports test

INTERVENTIONS:
Diagnostic Test: Return to sports test — The return-to-sport-tests are based on validated procedures commonly used in sports orthopedics, particularly following the stepwise testing concept described.
  Initially, the participant's individual sport level is determined via structured anamnesis. This is then followed by level-specific functional testing. Participants who do not perform Level 1 testing correctly will not proceed to Level 2 testing-even if their anamnesis suggests a higher sport level. This stepwise approach ensures safety and prevents injury during the testing process.

SUMMARY:
The ability to return to sports after joint arthroplasty is increasingly becoming an important factor for patients in terms of their perceived quality of life. In sports orthopaedics, standardized functional tests have already been established - particularly for anterior cruciate ligament injuries - to assess athletic performance and prevent re-injury. These tests allow a stepwise evaluation of a subject's physical readiness for sports.

In the field of arthroplasty, and despite increasing sports activity among patients with joint arthroplasty such structured assessment is still lacking. As a result, patients with arthroplasty typically resume sports activities based solely on individual recommendations from the surgeon or treating therapist. However, an objective evaluation of sports capability is currently not available.

Therefore the amendment intends to expand the current testing protocol of the already registered and ongoing study (Protocol ID: UBonn_TKA_FollowUp) to include additional standardized, evidence-based return-to-sprort-tests.

DETAILED DESCRIPTION:
These return-to-sports-tests are based on validated procedures commonly used in sports orthopaedics, particularly following the stepwise testing concept described by Keller et al..

Initially, the participant's individual sport level is determined via structured anamnesis. This is then followed by level-specific functional testing. Participants who do not perform Level 1 testing correctly will not proceed to Level 2 testing -even if their anamnesis suggests a higher sport level. This stepwise approach ensures safety and prevents injury during the testing process.

ELIGIBILITY:
Inclusion Criteria:

* The study includes all patients with a history of unicondylar or bicondylar knee joint replacement and engagement in sports activity.
* All participating patients have provided their informed consent following comprehensive information and explanation.
* All participating patients have signed the informed consent form for study participation as well as the data protection declaration after receiving detailed information and clarification.

Exclusion Criteria:

* Patients who are unable to understand the patient information and study design (e.g., due to language barriers) or whose compliance is deemed insufficient by the study team
* No knee joint endoprosthesis implanted
* No engagement in athletic activity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Level of sports 1-4 | Baseline at the time of measurement
  Levels of sports are divided into four levels:
  1. Sports without jumping;
  2. Dynamic sports without pivoting or abrupt stopping movements;
  3. Sports involving lateral movements and moderate pivoting or stopping motions (less intense than in Level 4);
  4. Sports with jumping, rapid pivoting, and sudden stopping movements.

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger von Eisenhart-Rothe, Univ. Prof. Dr. med., Study Chair — Department of Orthopaedics and Sports Orthopaedics
Locations (1):
- Department of Orthopaedics and Sports Orthopaedics, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The assessment regarding IPD with our data protection officer in relation to German and European data protection law has not yet been completed.

REFERENCES:
- [Background] Keller M, Kurz E, Schmidtlein O, Welsch G, Anders C. [Interdisciplinary Assessment Criteria for Rehabilitation after Injuries of the Lower Extremity: A Function-Based Return to Activity Algorithm]. Sportverletz Sportschaden. 2016 Mar;30(1):38-49. doi: 10.1055/s-0042-100966. Epub 2016 Mar 22. German. PMID 27002707